CLINICAL TRIAL: NCT02447185
Title: 25-Gauge Vitrectomy With Ranibizumab or Triamcinolone Acetonide on Proliferative Diabetic Retinopathy in China: a Randomized, Single Blind Trial
Brief Title: 25-G Vitrectomy With Ranibizumab or Triamcinolone Acetonide on PDR in China-Randomized Clinical Trial
Acronym: aiRTo-PDR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JUNYAN ZHANG (Other)
Collaborators: The First People's Hospital of Xuzhou (Other)
Responsible Party: Sponsor-Investigator, JUNYAN ZHANG, Senior Consultant and Statistician, The First People's Hospital of Xuzhou
Organization: The First People's Hospital of Xuzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PDR-RAN-RCT-LSY
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Lucentis; Ranibizumab; Triamcinolone Acetonide; Vitrectomy; PDR; 25-Gauge Vitrectomy
MeSH Terms: interventions — Ranibizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Experimental): A week before 25-gauge vitrectomy, all subjects in Ranibizumab group will receive Ranibizumab 0.5mg/0.05 ml intravitreal injection.
  During operation all subjects in this group will be injected Triamcinolone Acetonide 4 mg/0.1ml.
  All subjects in this group will get Ranibizumab 0.2 mg/0.02 ml intravitreal injection just after the operation.
  Interventions: Drug: Ranibizumab; Drug: Triamcinolone Acetonide
- Triamcinolone Acetonide (Active Comparator): A week before 25-gauge vitrectomy, all subjects in Triamcinolone Acetonide group will receive Triamcinolone Acetonide 4mg/0.1 ml intravitreal injection.
  During operation all subjects in this group will be injected Triamcinolone Acetonide 4 mg/0.1ml.
  All subjects in this group will get Triamcinolone Acetonide 1mg/0.025 ml intravitreal injection just after the operation.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Ranibizumab — A week before 25-gauge vitrectomy, all subjects in Ranibizumab group will receive Ranibizumab 0.5mg/0.05 ml intravitreal injection.
  All subjects in Ranibizumab group will get Ranibizumab 0.2 mg/0.02 ml intravitreal injection just after the operation.
  Other Names: rhuFab V2; Lucentis
  Arms: Ranibizumab
Drug: Triamcinolone Acetonide — A week before 25-gauge vitrectomy, all subjects in TA group will receive Triamcinolone Acetonide 4mg/0.1ml intravitreal injection.
  During operation all subjects in Ranibizumab group and in TA group will be injected Triamcinolone Acetonide 4 mg/0.1ml.
  All subjects in TA group will get Triamcinolone Acetonide 1mg/0.025 ml intravitreal injection just after the operation.
  Other Names: Vitreal S; Cinonide; Tricort 40; Kenalog

SUMMARY:
Proliferative diabetic retinopathy(PDR) is the leading cause of visual loss in diabetic patients. Operation is an efficient method to treat PDR. Anti-vascular endothelial growth factor (anti-VEGF) can be used as an adjuvant therapy which can make operation more easy.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy(PDR) is the leading cause of visual loss in diabetic patients. The operation indication includes non-absorbed vitreous haemorrhage, dense bleeding in front of the macular, proliferative vitreoretinopathy traction macular, tractional retinal detachment combined break, severe progressive fiber vascular proliferation and vitreous haemorrhage combined with early iris neovascularization.

Due to VEGF levels rise in vitreous cavity of PDR patients, some inflammatory cytokines involved in, make easy bleeding during surgery and heavier inflammatory reaction postoperation,thus affecting the curative effect of the operation.

Ranibizumab as angiogenesis inhibitors, has widely applied in the treatment of age-related macular degeneration, won the recognition of ophthalmologists.

Some scholars try to expand the application in diabetic macular edema, also obtained the good curative effect.Some scholars also applied the angiogenesis inhibitors to the diabetes retinopathy before surgery in the hope to reduce the occurrence of intraoperative bleeding.Compared with bevacizumab, the short half-life of lucentis, and thus reduce the inhibition of VEGF system risk.

In this project, the investigators will inject lucentis into vitreous cavity before surgery of PDR, and observe the effect and complications of the operation, compared with triamcinolone acetonide group(the control group); At the same time the cytokines level of VEGF, pigment epithelium-derived factor (PEDF), epidermal growth factor (EGF), Transforming Growth Factor-beta (TGF-beta), interleukin 6 (IL - 6) and interleukin 8 (IL - 8) will be detected before and after pretreatment with lucentis or triamcinolone acetonide, and the cytokines concentration change will be compared between two groups, the mechanism of PDR will be further clarified and theoretical basis for looking for treatment strategies will be a set.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus with Diabetic Retinopathy
* Vitreous hemorrhage/Proliferation of retinal/Tractional detachment of retina

Exclusion Criteria:

* Fasting blood-glucose more than 8mmol/ml
* Subjects who have operation on vitreous before
* Accompany with other ophthalmology diseases except cataract
* History of vitrectomy surgery in the study eye
* Previous subfoveal focal laser photocoagulation in the study eye
* Previous participation in a clinical trial (for either eye)
* Previous subfoveal focal laser photocoagulation in the study eye
* Other diseases cannot afford Vitrectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
intraoperative bleeding | during operation of 25-G Vitrectomy

SECONDARY OUTCOMES:
composite outcomes including amotio retinae,vitreous hemorrhage within 12 months after vitrectomy | 12 months after the last subject accepts vitrectomy
the change of Best-corrected visual acuity | the change of best-corrected visual acuity at month 12 after vitrectomy
the change of inflammatory factors in vitreous body | 7 days after the first injection

CONTACTS AND LOCATIONS:
Overall Officials: SUYAN LI, MD, Principal Investigator — Ophthalmology Department of the 1st People Hospital of Xuzhou
Locations (1):
- The First People Hospital of Xuzhou, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guthoff R, Riederle H, Meinhardt B, Goebel W. Subclinical choroidal detachment at sclerotomy sites after 23-gauge vitrectomy: analysis by anterior segment optical coherence tomography. Ophthalmologica. 2010;224(5):301-7. doi: 10.1159/000298750. Epub 2010 Mar 23. PMID 20332654
- [Result] Dehghan MH, Salehipour M, Naghib J, Babaeian M, Karimi S, Yaseri M. Pars plana vitrectomy with internal limiting membrane peeling for refractory diffuse diabetic macular edema. J Ophthalmic Vis Res. 2010 Jul;5(3):162-7. PMID 22737351
- [Result] Cho M, D'Amico DJ. Transconjunctival 25-gauge pars plana vitrectomy and internal limiting membrane peeling for chronic macular edema. Clin Ophthalmol. 2012;6:981-9. doi: 10.2147/OPTH.S33391. Epub 2012 Jul 6. PMID 22848140
- [Result] Song SJ, Sohn JH, Park KH. Evaluation of the efficacy of vitrectomy for persistent diabetic macular edema and associated factors predicting outcome. Korean J Ophthalmol. 2007 Sep;21(3):146-50. doi: 10.3341/kjo.2007.21.3.146. PMID 17804919
- [Result] Gupta V, Arevalo JF. Surgical management of diabetic retinopathy. Middle East Afr J Ophthalmol. 2013 Oct-Dec;20(4):283-92. doi: 10.4103/0974-9233.120003. PMID 24339677
- [Result] Shamsi HN, Masaud JS, Ghazi NG. Diabetic macular edema: New promising therapies. World J Diabetes. 2013 Dec 15;4(6):324-38. doi: 10.4239/wjd.v4.i6.324. PMID 24379924
- [Result] Romero-Aroca P. Managing diabetic macular edema: The leading cause of diabetes blindness. World J Diabetes. 2011 Jun 15;2(6):98-104. doi: 10.4239/wjd.v2.i6.98. PMID 21860693
- [Result] Bainbridge J. Refractory diabetic macular edema. J Ophthalmic Vis Res. 2010 Jul;5(3):143-4. No abstract available. PMID 22737347
- [Result] Jahn CE, Topfner von Schutz K, Richter J, Boller J, Kron M. Improvement of visual acuity in eyes with diabetic macular edema after treatment with pars plana vitrectomy. Ophthalmologica. 2004 Nov-Dec;218(6):378-84. doi: 10.1159/000080940. PMID 15564755
- [Result] Robaszkiewicz J, Chmielewska K, Wierzbowska J, Figurska M, Frontczak-Baniewicz M, Stankiewicz A. [Combined surgical and pharmacological treatment of diabetic maculopathy]. Klin Oczna. 2010;112(1-3):19-23. Polish. PMID 20572497